CLINICAL TRIAL: NCT01362959
Title: Nicotine Replacement Therapy in the Intensive Care Unit: a Randomized, Controlled Pilot Study
Brief Title: Nicotine Replacement Therapy in the Intensive Care Unit
Acronym: NicGoWell
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gelderse Vallei Hospital (Other)
Collaborators: Deventer Ziekenhuis (Other); Wageningen University (Other)
Responsible Party: Principal Investigator, drs. B. de Jong, MD, Gelderse Vallei Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NicGoWell1.0; 2011-002458-29 (EudraCT Number)
Record Dates: First submitted 2011-05-26; First posted 2011-06-01 (Estimated); Results first posted 2018-10-10 (Actual); Last update posted 2018-10-10 (Actual); Status verified 2018-03

CONDITIONS: Delirium; Psychomotor Agitation; Substance Withdrawal Syndrome; Nicotine Replacement Therapy
Keywords: Delirium; Psychomotor Agitation; Substance Withdrawal Syndrome; Nicotine replacement therapy
MeSH Terms: conditions — Delirium; Psychomotor Agitation; Substance Withdrawal Syndrome | interventions — Tobacco Use Cessation Devices; Transdermal Patch

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nicotine patch (Experimental)
  Interventions: Drug: Transdermal nicotine patch
- Control patch (Placebo Comparator): The control product is a look-alike patch compared to the test product, containing no nicotine or other active substances.
  Interventions: Other: Cutaneous patch, containing no active substances

INTERVENTIONS:
Drug: Transdermal nicotine patch — The test product is a transdermal nicotine patch. The dosage of the test product depends on the amount of cigarettes used by a specific patient (21 or more or less than 21) delivering 21 or 14 mg nicotine/24 hrs. During the study period of thirty (30) days a patch will be applicated daily.
  Other Names: Nicotinell patch, regulated delivery 35 mg. RVG 14830; Nicotinell patch, regulated delivery 52.5 mg. RVG 14831
  Arms: Nicotine patch
Other: Cutaneous patch, containing no active substances — During the study period of thirty (30) days, the control product will be applicated daily.
  Arms: Control patch

SUMMARY:
The purpose of this study is to determine whether transdermal nicotine replacement therapy is safe and effective for treating nicotine withdrawal symptoms in the critically ill smoking patient.

DETAILED DESCRIPTION:
Cigarette smoking remains the leading cause of preventable disease and premature death worldwide. There are about 1.2 billion smokers in the world, half of whom will die from diseases caused by smoking. Smoking causes 5 million deaths per year, and if present trends continue, 10 million smokers per year are projected to die by 2025.

Furthermore, abstinence from the highly addictive tobacco products can lead to withdrawal symptoms. Although these symptoms are non-life threatening in healthy and hospitalized adults they are not well described in the mechanically ventilated active smoking patient.

Retrospective studies found a higher, lower or equal mortality in critically ill patients receiving nicotine replacement therapy compared to patients receiving no nicotine replacement.

Because of these conflicting results and the absence of a randomized controlled trial studying the efficacy and safety of transdermal nicotine replacement therapy in the critically ill smoking patient a clinical study will be conducted.

ELIGIBILITY:
Inclusion Criteria: Any patient admitted to the intensive care unit must meet all of the following criteria to be eligible for the study:

* Critically ill active smoking patient
* Being mechanically ventilated
* Start of study product application within 48 hours after ICU admission
* Expected to be mechanically ventilated for more than 48 hours after start of application of the study product

Exclusion Criteria: Any patient admitted to the intensive care unit meeting one or more of the following criteria is not eligible for the study:

* Patient younger than 18 years
* Patient or next of kin denying research authorization
* Pregnancy
* Breastfeeding women
* History of chronic dementia or psychosis
* (Acute) neurologic disease on admission, possibly confounding study objectives (TBI, stroke, ICH/SAH, seizures, meningitis, encephalitis, intracranial tumor)
* Patient receiving any form of NRT within two weeks before admission
* Patient not understanding Dutch
* Patient with acute myocardial infarction
* Patient with severe cardiac arrhythmia
* Patient with unstable or deteriorating angina pectoris
* Patient with generalized acute or chronic skin diseases interfering with NRT absorption
* Patient with severe hearing deficiency
* Moribund patient
* Patient with known hypersensibility to nicotine or components of the transdermal therapeutic system
* Patient with known hypersensibility to patches
* Patient participating in an other study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2012-06; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ben Jong,de, MD, Principal Investigator — Gelderse Vallei Hospital
Locations (2):
- Netherlands (2):
  - Gelderse Vallei Hospital, Ede, Gelderland
  - Deventer Hospital, Deventer, Overijssel

REFERENCES:
- [Background] Hays JT, Ebbert JO. Adverse effects and tolerability of medications for the treatment of tobacco use and dependence. Drugs. 2010 Dec 24;70(18):2357-72. doi: 10.2165/11538190-000000000-00000. PMID 21142259
- [Background] Moss M, Burnham EL. Alcohol abuse in the critically ill patient. Lancet. 2006 Dec 23;368(9554):2231-42. doi: 10.1016/S0140-6736(06)69490-7. PMID 17189035
- [Background] Benowitz NL. Nicotine addiction. N Engl J Med. 2010 Jun 17;362(24):2295-303. doi: 10.1056/NEJMra0809890. No abstract available. PMID 20554984
- [Background] Hatsukami DK, Stead LF, Gupta PC. Tobacco addiction. Lancet. 2008 Jun 14;371(9629):2027-38. doi: 10.1016/S0140-6736(08)60871-5. PMID 18555914
- [Background] Mills EJ, Wu P, Lockhart I, Wilson K, Ebbert JO. Adverse events associated with nicotine replacement therapy (NRT) for smoking cessation. A systematic review and meta-analysis of one hundred and twenty studies involving 177,390 individuals. Tob Induc Dis. 2010 Jul 13;8(1):8. doi: 10.1186/1617-9625-8-8. PMID 20626883
- [Background] Lucidarme O, Seguin A, Daubin C, Ramakers M, Terzi N, Beck P, Charbonneau P, du Cheyron D. Nicotine withdrawal and agitation in ventilated critically ill patients. Crit Care. 2010;14(2):R58. doi: 10.1186/cc8954. Epub 2010 Apr 9. PMID 20380688
- [Background] Mayer SA, Chong JY, Ridgway E, Min KC, Commichau C, Bernardini GL. Delirium from nicotine withdrawal in neuro-ICU patients. Neurology. 2001 Aug 14;57(3):551-3. doi: 10.1212/wnl.57.3.551. PMID 11502936
- [Background] Moreno R, Vincent JL, Matos R, Mendonca A, Cantraine F, Thijs L, Takala J, Sprung C, Antonelli M, Bruining H, Willatts S. The use of maximum SOFA score to quantify organ dysfunction/failure in intensive care. Results of a prospective, multicentre study. Working Group on Sepsis related Problems of the ESICM. Intensive Care Med. 1999 Jul;25(7):686-96. doi: 10.1007/s001340050931. PMID 10470572
- [Background] Lee AH, Afessa B. The association of nicotine replacement therapy with mortality in a medical intensive care unit. Crit Care Med. 2007 Jun;35(6):1517-21. doi: 10.1097/01.CCM.0000266537.86437.38. PMID 17452926
- [Background] Paciullo CA, Short MR, Steinke DT, Jennings HR. Impact of nicotine replacement therapy on postoperative mortality following coronary artery bypass graft surgery. Ann Pharmacother. 2009 Jul;43(7):1197-202. doi: 10.1345/aph.1L423. Epub 2009 Jun 30. PMID 19567657
- [Background] Seder DB, Schmidt JM, Badjatia N, Fernandez L, Rincon F, Claassen J, Gordon E, Carrera E, Kurtz P, Lee K, Connolly ES, Mayer SA. Transdermal nicotine replacement therapy in cigarette smokers with acute subarachnoid hemorrhage. Neurocrit Care. 2011 Feb;14(1):77-83. doi: 10.1007/s12028-010-9456-9. PMID 20949331
- [Background] Cartin-Ceba R, Warner DO, Hays JT, Afessa B. Nicotine replacement therapy in critically ill patients: a prospective observational cohort study. Crit Care Med. 2011 Jul;39(7):1635-40. doi: 10.1097/CCM.0b013e31821867b8. PMID 21494111
- [Background] Horan TC, Andrus M, Dudeck MA. CDC/NHSN surveillance definition of health care-associated infection and criteria for specific types of infections in the acute care setting. Am J Infect Control. 2008 Jun;36(5):309-32. doi: 10.1016/j.ajic.2008.03.002. No abstract available. PMID 18538699
- [Background] Centers for Disease Control and Prevention (CDC). Vital signs: central line-associated blood stream infections--United States, 2001, 2008, and 2009. MMWR Morb Mortal Wkly Rep. 2011 Mar 4;60(8):243-8. PMID 21368740
- [Background] Hsieh SJ, Ware LB, Eisner MD, Yu L, Jacob P 3rd, Havel C, Goniewicz ML, Matthay MA, Benowitz NL, Calfee CS. Biomarkers increase detection of active smoking and secondhand smoke exposure in critically ill patients. Crit Care Med. 2011 Jan;39(1):40-5. doi: 10.1097/CCM.0b013e3181fa4196. PMID 20935560
- [Derived] de Jong B, Schuppers AS, Kruisdijk-Gerritsen A, Arbouw MEL, van den Oever HLA, van Zanten ARH. The safety and efficacy of nicotine replacement therapy in the intensive care unit: a randomised controlled pilot study. Ann Intensive Care. 2018 Jun 7;8(1):70. doi: 10.1186/s13613-018-0399-1. PMID 29881956
- See also: Website Gelderse Vallei Hospital — http://www.geldersevallei.nl

RESULTS

PARTICIPANT FLOW:
Groups:
- Nicotine Patch: Transdermal nicotine patch: The test product is a transdermal nicotine patch. The dose of the test product depends on the amount of cigarettes used by a specific patient (21 or more or less than 21) delivering 21 or 14 mg nicotine/24 hrs. During the study period of thirty (30) days a patch will be applied daily.
- Control Patch: The control product is a look-alike cutaneous patch comparable to the test product, containing no nicotine or other active substances. During the study period of thirty (30) days, the control product will be applied daily.
Period: Overall Study
Arm/Group | Nicotine Patch | Control Patch
Started | 21 | 26
Completed | 21 | 26
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Nicotine Patch: Transdermal nicotine patch: The test product is a transdermal nicotine patch. The dosage of the test product depends on the amount of cigarettes used by a specific patient (21 or more or less than 21) delivering 21 or 14 mg nicotine/24 hrs. During the study period of thirty (30) days a patch will be applied daily.
- Total: Total of all reporting groups
Arm/Group | Nicotine Patch | Control Patch | Total
Number analyzed (Participants) | 21 | 26 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] — Years
  years | 60.1 (10.55) | 65.2 (9.13) | 62.9 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 19
  Male | 12 | 16 | 28
Region of Enrollment [Number; unit: participants]
  Netherlands | 21 | 26 | 47

OUTCOME MEASURES:

1. Primary Outcome: 30-day Mortality
Time Frame: 30 days
Measure: Number; unit: percentage of patients
Arm/Group | Nicotine Replacement | Control
Number analyzed (Participants) | 21 | 26
percentage of patients | 9.5 | 7.7

2. Primary Outcome: Patient Location Day 30
Description: In the ICU or hospital at day 30
Time Frame: On day 30
Measure: Count of Participants; unit: Participants
Arm/Group | Nicotine Replacement | Control
Number analyzed (Participants) | 21 | 26
Participants | 1 | 11

3. Secondary Outcome: 90-day Mortality
Description: Mortality at day 90 after enrollment
Time Frame: Day 90 followup
Measure: Number; unit: percentage of patients
Arm/Group | Nicotine Replacement | Control
Number analyzed (Participants) | 21 | 26
percentage of patients | 14.3 | 19.2

4. Post Hoc Outcome: Time in Normal Brain Function D20
Description: Time spent alive without delirium and without sedation or coma
Time Frame: 20 days
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Nicotine Replacement | Control
Number analyzed (Participants) | 21 | 26
hours | 400 [316 to 448] | 304 [110 to 432]

5. Post Hoc Outcome: Time in Normal Brain Function D10
Description: Time alive without delirium and without sedation or coma
Time Frame: 10 days
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Nicotine Replacement | Control
Number analyzed (Participants) | 21 | 26
hours | 160 [96 to 216] | 88 [20 to 210]

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Nicotine Replacement | Control
All-Cause Mortality (participants affected / at risk) | 2/21 | 2/26
Serious Adverse Events (participants affected / at risk) | 4/21 | 11/26
Other Adverse Events (participants affected / at risk) | 21/21 | 26/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nicotine Replacement (N=21) | Control (N=26)
Death due to respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) — Respiratory failure, hypoxaemia
Death due to hypercapnic coma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Hypercarbia due to type II respiratory failure
Hemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Blood in the thoracic cavity
Reintubation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) — Need for reintubation after extubation
Death due to septic shock (Infections and infestations) | 0 (0) | 1 (1) — Respiratory sepsis, leading to death
haemorrhagic shock (Vascular disorders) | 0 (0) | 1 (1) — Shock due to severe hemorrhage
Stoma necrosis (Gastrointestinal disorders) | 0 (0) | 1 (1) — Necrosis of colostoma
Duodenal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) — Perforation of duodenum
Ischaemic colitis (Gastrointestinal disorders) | 0 (0) | 2 (2) — Ischaemic disease of colon
Asystole (Cardiac disorders) | 0 (0) | 1 (1) — Absence of cardiac rhythm
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nicotine Replacement (N=21) | Control (N=26)
Electrolyte disturbance (Investigations) | 21 (36) | 26 (49) — Any type of electrolyte distubance
Gastrointestinal event (Gastrointestinal disorders) | 21 (27) | 26 (40) — Any type of gastrointestinal upset
Cardiovascular (Cardiac disorders) | 16 (16) | 26 (43) — Any type of cardiac or circulatory event
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 8 (8) — Any type of pulmonary event
Renal (Renal and urinary disorders) | 1 (1) | 6 (6) — Any type of renal disorder
Other adverse events (General disorders) | 17 (17) | 26 (31) — Any other type of adverse event

LIMITATIONS AND CAVEATS:
Pilot study, therefore small numbers

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No